CLINICAL TRIAL: NCT01996397
Title: Acute Feedback on Left ventrIcular Lead Implantation Location for Cardiac Resynchronization Therapy
Acronym: CCI impact
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Principal Investigator, Erik Kongsgaard, MD, Ph.d, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2013/140
Record Dates: First submitted 2013-11-01; First posted 2013-11-27 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Heart Failure; Resynchronization Therapy; Assessment of Acute CRT Response
Keywords: Heart failure; Bundle branch block; CRT response
MeSH Terms: conditions — Heart Failure; Bundle-Branch Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CRT implantation (Other): Standard CRT indication. Assessment of acute response to CRT.
  Interventions: Procedure: Cardiac resynchronization therapy device implantation

INTERVENTIONS:
Procedure: Cardiac resynchronization therapy device implantation

SUMMARY:
Exploratory, prospective, interventional, non-randomized single-center research study to compare metrics derived from 2 or 3-D reconstructions of lead movement, bioimpedance and VCG to augmentation of left ventricular contractility (LV dP/dt max) at different pacing configurations in patients undergoing a CRT-implant. Pacing sites and contractility data will be compared to pre operative cardiac ultrasound and MRI metrics.

ELIGIBILITY:
Inclusion Criteria:

* Subject is indicated for CRT or CRT-D device according to current applicable ESC/AHA guidelines
* Subject is in stable sinus rhythm at the time of implant (no atrial arrhythmias lasting > 30 seconds during the last 2 weeks prior to inclusion). No documented AF-episodes allowed during the last 2 weeks prior to inclusion.
* Subject receives optimal heart failure oral medical therapy (ACE inhibitor and/or ARB and Beta Blockers), and is on a stable medication scheme for at least 2 months prior to enrollment.
* Subject (or the legal guardian) is willing to sign informed consent form

Exclusion Criteria:

* Permanent atrial fibrillation/ flutter or tachycardia
* RBBB
* Recent myocardial infarction (MI), within 40 days prior to enrollment. Subject underwent coronary artery bypass graft (CABG) or valve surgery, within 90 days prior to enrollment
* Post heart transplantation, or is actively listed on the transplantation list, or has reasonable probability (per investigator's discretion) of undergoing transplantation in the next year
* Implanted with a left ventricular assist device (LVAD), or has reasonable probability (per investigator's discretion) of receiving a LVAD in the next year
* On chronic renal dialysis, or with severe renal disease (defined as estimated Glomerular Filtration Rate (equation provided by Modification of Diet in Renal Disease study): (eGFR) < 30 mL/min/1.73m2)
* On continuous or uninterrupted infusion (inotropic) therapy for heart failure (≥ 2 stable infusions a week)
* Severe aortic stenosis (with a valve area of <1.0 cm2 or significant valve disease expected to be operated on within study period)
* Complex and uncorrected congenital heart disease
* Mechanical heart valve
* Breastfeeding women, or women of child bearing potential and who are not on a reliable form of birth control
* Enrolled in one or more concurrent studies that would confound the results of this study
* Already implanted with pacemaker (CRT, CRT-D, ICD) and needs replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
dP\dt max response to different ventricular lead pacing sites | 6 months
  To compare metrics derived from 2 or 3-D reconstructions of lead movement to augmentation of left ventricular contractility (LV dP/dt max) at different pacing configurations in patients undergoing a CRT-implant Main objective is to identify the optimal LV pacing site within each patient where the force of contraction during BiV pacing is maximized and to assess the feasibility of a non-invasive sensor to identify this optimal site.

SECONDARY OUTCOMES:
Lead movements and electrical measures | 6 months
  Compare metrics derived from 2/3-D reconstructions of lead movement to electrical measures (e.g. Q-LV-timing or VCG) at different pacing configurations in patients undergoing a CRT-implant.
Metrics derived from 2/3-D reconstructions of lead movement and Force-Interval-Relation | 6 months
  To compare metrics derived from 2/3-D reconstructions of lead movement to Force-Interval-Relation at different pacing configurations in patients undergoing a CRT-implant.
Metrics derived from 2/3-D reconstructions of lead movement and CardioGuide Motion Map | 6 months
  To compare metrics derived from 2/3-D reconstructions of lead movement to CardioGuide Motion Map at different pacing configurations in patients undergoing a CRT-implant.

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Rikshospitalet, Oslo, Oslo County, Norway

REFERENCES:
- [Background] Bristow MR, Saxon LA, Boehmer J, Krueger S, Kass DA, De Marco T, Carson P, DiCarlo L, DeMets D, White BG, DeVries DW, Feldman AM; Comparison of Medical Therapy, Pacing, and Defibrillation in Heart Failure (COMPANION) Investigators. Cardiac-resynchronization therapy with or without an implantable defibrillator in advanced chronic heart failure. N Engl J Med. 2004 May 20;350(21):2140-50. doi: 10.1056/NEJMoa032423. PMID 15152059
- [Background] Cleland JG, Daubert JC, Erdmann E, Freemantle N, Gras D, Kappenberger L, Tavazzi L; Cardiac Resynchronization-Heart Failure (CARE-HF) Study Investigators. The effect of cardiac resynchronization on morbidity and mortality in heart failure. N Engl J Med. 2005 Apr 14;352(15):1539-49. doi: 10.1056/NEJMoa050496. Epub 2005 Mar 7. PMID 15753115
- [Background] Abraham WT, Fisher WG, Smith AL, Delurgio DB, Leon AR, Loh E, Kocovic DZ, Packer M, Clavell AL, Hayes DL, Ellestad M, Trupp RJ, Underwood J, Pickering F, Truex C, McAtee P, Messenger J; MIRACLE Study Group. Multicenter InSync Randomized Clinical Evaluation. Cardiac resynchronization in chronic heart failure. N Engl J Med. 2002 Jun 13;346(24):1845-53. doi: 10.1056/NEJMoa013168. PMID 12063368
- [Background] Fornwalt BK, Sprague WW, BeDell P, Suever JD, Gerritse B, Merlino JD, Fyfe DA, Leon AR, Oshinski JN. Agreement is poor among current criteria used to define response to cardiac resynchronization therapy. Circulation. 2010 May 11;121(18):1985-91. doi: 10.1161/CIRCULATIONAHA.109.910778. Epub 2010 Apr 26. PMID 20421518
- [Background] Butter C, Auricchio A, Stellbrink C, Fleck E, Ding J, Yu Y, Huvelle E, Spinelli J; Pacing Therapy for Chronic Heart Failure II Study Group. Effect of resynchronization therapy stimulation site on the systolic function of heart failure patients. Circulation. 2001 Dec 18;104(25):3026-9. doi: 10.1161/hc5001.102229. PMID 11748094
- [Background] Rossillo A, Verma A, Saad EB, Corrado A, Gasparini G, Marrouche NF, Golshayan AR, McCurdy R, Bhargava M, Khaykin Y, Burkhardt JD, Martin DO, Wilkoff BL, Saliba WI, Schweikert RA, Raviele A, Natale A. Impact of coronary sinus lead position on biventricular pacing: mortality and echocardiographic evaluation during long-term follow-up. J Cardiovasc Electrophysiol. 2004 Oct;15(10):1120-5. doi: 10.1046/j.1540-8167.2004.04089.x. PMID 15485432
- [Background] Merchant FM, Heist EK, McCarty D, Kumar P, Das S, Blendea D, Ellinor PT, Mela T, Picard MH, Ruskin JN, Singh JP. Impact of segmental left ventricle lead position on cardiac resynchronization therapy outcomes. Heart Rhythm. 2010 May;7(5):639-44. doi: 10.1016/j.hrthm.2010.01.035. Epub 2010 Feb 1. PMID 20298819
- [Background] Mullens W, Verga T, Grimm RA, Starling RC, Wilkoff BL, Tang WHW. Persistent hemodynamic benefits of cardiac resynchronization therapy with disease progression in advanced heart failure. J Am Coll Cardiol. 2009 Feb 17;53(7):600-607. doi: 10.1016/j.jacc.2008.08.079. PMID 19215835
- [Background] Blendea D, Singh JP. Lead positioning strategies to enhance response to cardiac resynchronization therapy. Heart Fail Rev. 2011 May;16(3):291-303. doi: 10.1007/s10741-010-9212-4. PMID 21184174
- [Background] Duckett SG, Ginks M, Shetty AK, Bostock J, Gill JS, Hamid S, Kapetanakis S, Cunliffe E, Razavi R, Carr-White G, Rinaldi CA. Invasive acute hemodynamic response to guide left ventricular lead implantation predicts chronic remodeling in patients undergoing cardiac resynchronization therapy. J Am Coll Cardiol. 2011 Sep 6;58(11):1128-36. doi: 10.1016/j.jacc.2011.04.042. PMID 21884950
- [Background] Bogaard MD, Houthuizen P, Bracke FA, Doevendans PA, Prinzen FW, Meine M, van Gelder BM. Baseline left ventricular dP/dtmax rather than the acute improvement in dP/dtmax predicts clinical outcome in patients with cardiac resynchronization therapy. Eur J Heart Fail. 2011 Oct;13(10):1126-32. doi: 10.1093/eurjhf/hfr094. Epub 2011 Jul 26. PMID 21791536
- [Background] Butter C, Stellbrink C, Belalcazar A, Villalta D, Schlegl M, Sinha A, Cuesta F, Reister C. Cardiac resynchronization therapy optimization by finger plethysmography. Heart Rhythm. 2004 Nov;1(5):568-75. doi: 10.1016/j.hrthm.2004.07.002. PMID 15851221
- [Background] Whinnett ZI, Davies JE, Willson K, Chow AW, Foale RA, Davies DW, Hughes AD, Francis DP, Mayet J. Determination of optimal atrioventricular delay for cardiac resynchronization therapy using acute non-invasive blood pressure. Europace. 2006 May;8(5):358-66. doi: 10.1093/europace/eul017. PMID 16635996
- [Background] Whinnett ZI, Davies JE, Willson K, Manisty CH, Chow AW, Foale RA, Davies DW, Hughes AD, Mayet J, Francis DP. Haemodynamic effects of changes in atrioventricular and interventricular delay in cardiac resynchronisation therapy show a consistent pattern: analysis of shape, magnitude and relative importance of atrioventricular and interventricular delay. Heart. 2006 Nov;92(11):1628-34. doi: 10.1136/hrt.2005.080721. Epub 2006 May 18. PMID 16709698
- [Background] Bocchiardo M, Meyer zu Vilsendorf D, Militello C, Lippert M, Czygan G, Schauerte P, Gaita F, Stellbrink C. Resynchronization therapy optimization by intracardiac impedance. Europace. 2010 Nov;12(11):1589-95. doi: 10.1093/europace/euq273. Epub 2010 Jul 28. PMID 20667892
- [Background] Turcott RG, Witteles RM, Wang PJ, Vagelos RH, Fowler MB, Ashley EA. Measurement precision in the optimization of cardiac resynchronization therapy. Circ Heart Fail. 2010 May;3(3):395-404. doi: 10.1161/CIRCHEARTFAILURE.109.900076. Epub 2010 Feb 22. PMID 20176716
- [Background] Jia P, Ramanathan C, Ghanem RN, Ryu K, Varma N, Rudy Y. Electrocardiographic imaging of cardiac resynchronization therapy in heart failure: observation of variable electrophysiologic responses. Heart Rhythm. 2006 Mar;3(3):296-310. doi: 10.1016/j.hrthm.2005.11.025. PMID 16500302
- [Background] Shetty AK, Duckett SG, Ma YL, Kapetanakis S, Ginks M, Bostock J, Carr-White G, Rhode K, Razavi R, Rinaldi CA. The acute hemodynamic response to LV pacing within individual branches of the coronary sinus using a quadripolar lead. Pacing Clin Electrophysiol. 2012 Feb;35(2):196-203. doi: 10.1111/j.1540-8159.2011.03268.x. Epub 2011 Nov 29. PMID 22126664
- [Background] Tysler M, Kneppo P, Turzova M, Svehlikova J, Karas S, Heblakova E, Hana K, Filipova S. Noninvasive assessment of local myocardium repolarization changes using high resolution surface ECG mapping. Physiol Res. 2007;56 Suppl 1:S133-S141. doi: 10.33549/physiolres.931312. Epub 2007 May 31. PMID 17552884
- [Background] van Deursen C, van Geldorp IE, Rademakers LM, van Hunnik A, Kuiper M, Klersy C, Auricchio A, Prinzen FW. Left ventricular endocardial pacing improves resynchronization therapy in canine left bundle-branch hearts. Circ Arrhythm Electrophysiol. 2009 Oct;2(5):580-7. doi: 10.1161/CIRCEP.108.846022. Epub 2009 Aug 10. PMID 19843927
- See also: Center for Cardiological Innovation — http://www.heart-sfi.no/
- See also: Oslo University Hospital — http://www.oslo-universitetssykehus.no